CLINICAL TRIAL: NCT02982135
Title: Direct Bypass Versus Indirect Bypass in Treatment of Adults Hemorrhagic Moyamoya Disease:a Prospective Multi-center Cohort Study
Brief Title: Direct Bypass Versus Indirect Bypass in Treatment of Adults Hemorrhagic Moyamoya Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: liuxingju (Other Government)
Responsible Party: Sponsor-Investigator, liuxingju, Principal investigator, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BJTTH-003
Record Dates: First submitted 2016-11-20; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Moyamoya Disease
Keywords: hemorrhagic moyamoya disease; bypass; indirect bypass
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 direct bypass (Other): direct bypass : patients recieve direct bypass treatment
  Interventions: Other: bypass surgery and indrect bypass surgery
- group 2 indirect bypass (Other): indirect bypass: patients recieve indirect bypass treatment
  Interventions: Other: bypass surgery and indrect bypass surgery

INTERVENTIONS:
Other: bypass surgery and indrect bypass surgery — bypass surgery ： patients recieved STA-MCA bypass indrect bypass surgery：patients recieved EDAS or mutiple bur holes

SUMMARY:
The investigators conducted a prospective multi-center study assessing the effect of direct bypass and indrect bypass in treatment of hemorrhagic moyamoya disease.

ELIGIBILITY:
Inclusion Criteria:

1. cerebral digital subtraction contrast angiography (DSA) revealed severe stenosis or occlusion of the distal internal carotid or proximal middle and anterior cerebral arteries with prominent lenticulostriate "moyamoya collaterals"
2. patients had experienced at least one intracranial hemorrhage which was verified by computed tomography (CT) scanning, magnetic resonance imaging MRI), or lumbar puncture.
3. Patients requiring surgery

Exclusion Criteria:

1. Patient whose initial onset was marked by ischemia but subsequently suffered from intracranial hemorrhage
2. patients refused to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
rebleeding events | 5-10 years

SECONDARY OUTCOMES:
ischemic events | 5-10 years
postoperative compilications | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes